CLINICAL TRIAL: NCT03665142
Title: Efficacy of Kinesio Taping on Pain, Pain Threshold and Emotional Status in Tension Type Headache
Brief Title: Efficacy of Kinesio Taping in Tension Type Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, TOMRIS DUYMAZ, Principal Investigator, Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBU2018
Record Dates: First submitted 2018-09-06; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Tension-Type Headache
Keywords: Tension-Type Headache; Kinesio Tape; Pain
MeSH Terms: conditions — Tension-Type Headache; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Patients were randomly divided into 2 groups. A randomized list is prepared in a computer environment by a statistician for randomization. In this list, the odd numbers for the control group and the KT group were given double numbers. The group identification is printed on sequentially numbered cards placed in sealed envelopes. After enrollment, the numbered envelope was opened by the patient and the blind investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio taping (Experimental): In this study, Kinesio Tape Tex Gold® kinesio tape over lateral ankle (5cm*5m) is used. 36 participants were taped for the TTH.50-mm wide and 0.5-mm thick KT was applied to the upper trapezius muscle with one I-shaped tape. The tape was measured from the acromion to the hairline at the back, and the upper trapezius fibers were extended in the extended position, ie the cervical vertebrae were flexed to the opposite side and applied to the same side in the flexion and rotation position.
  Interventions: Other: Kinesio taping
- Exercise (Placebo Comparator): Upper trapezius muscle stretching exercise was applied to the control group.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Kinesio taping — Upper trapezius muscle stretching exercise with Kinesio taping (KT) was applied to the study group. KT was applied 8 times in total for 4 weeks with 2 sessions per week. Stretching exercise was done in the morning, afternoon and evening 3 times (repeated 10 times per set) every day for 4 weeks and 5 days of the week.
  Arms: Kinesio taping
Other: Exercise — Upper trapezius muscle stretching exercise was applied to the control group.
  Arms: Exercise

SUMMARY:
Aim: The purpose of this study was to investigate the efficacy of Kinesio taping on upper trapezius muscle on the reduction of pain and emotional state in the treatment of patients with tension type headache by acting on myofacial mechanoreceptors.

Methods: This study was conducted in 71 patients aged 30-45 years with tension type headache diagnosed. Patients were randomly divided into 2 groups. While KT and stretching exercises were performed in the study group, only the stretching exercise was performed for the control group. KT was applied 8 times in total for 4 weeks with 2 sessions per week. Stretching exercise was done in the morning, afternoon and evening 3 times every day for 4 weeks and 5 days of the week. After recording the demographic data of all the patients participating in the study, assessed the sensitivity of the right and left upper parts of the trapezius with algometer, pain intensity with visual analog scale (VAS), Beck depression and anxiety scale for emotional status before and after treatment. p < 0.05 was considered statistically significant.

DETAILED DESCRIPTION:
Participants This study was performed with 71 patients diagnosed as tension type headache. The study was conducted with patients at the Florence Nightingale Hospital between the ages of 30-45 who applied to the Neurology clinic. Patients were randomly divided into 2 groups. A randomized list is prepared in a computer environment by a statistician for randomization. In this list, the odd numbers for the control group and the KT group were given double numbers. The group identification is printed on sequentially numbered cards placed in sealed envelopes. After enrollment, the numbered envelope was opened by the patient and the blind investigator. Patients were included in the study, between 30 and 45 years of age, who had a tension headache diagnosis, presence of a tender points on the upper part of the trapezoid, voluntary or written volunteers to participate in the study. Exclusion criteria include cervical area surgery and / or surgery, cervical trauma history, systemic disease targeting this area, moderate or excessive nausea and vomiting with headache, headache due to other causes (e.g., subarachnoid hemorrhage, cerebral hemorrhage, cerebral embolism, cerebral thrombosis, vascular malformation, arthritis, hypertension, or arteriosclerosis), have used prophylactic headache medications in the last 3 months, neurological, mental, hemorrhagic disease, allergy, serious heart, liver, kidney and other organ deficiencies.

Interventions Upper trapezius muscle stretching exercise with KT was applied to the study group, and upper trapezius muscle stretching exercise was applied to the control group. KT was applied 8 times in total for 4 weeks with 2 sessions per week. Stretching exercise was done in the morning, afternoon and evening 3 times (repeated 10 times per set) every day for 4 weeks and 5 days of the week.

KT application: 50-mm wide and 0.5-mm thick KT was applied to the upper trapezius muscle with one I-shaped tape. The tape was measured from the acromion to the hairline at the back, and the upper trapezius fibers were extended in the extended position, ie the cervical vertebrae were flexed to the opposite side and applied to the same side in the flexion and rotation position. The band was fixed to the insertion site of the acromion in the initial resting position. The muscle was lengthened and the band was fixed with the initial skin shift, then the band was fixed to the origin of the hairline from the muscle fixed with 10% stretch. The tape was rubbed together with the muscle in the extended position.

Outcome measurements After recording the demographic data of all the patients participating in the study, the sensitivity of the right and left upper parts of the trapezius assessed with algometer, pain intensity with visual analog scale (VAS), Beck depression and anxiety scale for emotional status before and after treatment.

The algometer is a mechanical pressure device with a minimum diameter of 100 g and a pressure of 10 kg / cm2, with a spring-loaded cylinder with a rubber tip, a circle and a pressure surface of 1 cm2 in diameter, obtained in kg / cm2. Before measuring with the algo- rithm, a pressure of approximately 4 kg was applied to the midpoint of the upper part of the trapezius muscle, which is the control point, with the pulp of the thumb of the hand. Then the force was applied to the same point, causing pain to separate the patient's sense of pressure and pain sensation. This process has been repeated several times. Measurements with an algometer were made at a rate of 1 kg per second. The measurements were interrupted for at least 15-20 seconds. Three measurements were made at these 2 sensitive points and the average of the measurements was recorded.

Visual Analog Scale (VAS) is used to convert some numerical values, such as pain, to numeric values. The two extremes of a 100 mm line are to be assessed on two extremes and the patient is asked to indicate on the line where the severity of the pain is appropriate by drawing a line or placing a point or pointing. The length of the distance from where the pain has never occurred to the point the patient has marked indicates the pain of the patient.

Beck Depression Inventory (BDI) and Beck Anxiety Inventory (BAI) developed by Aron T. Beck in 1961, Turkish validity and reliability were done by Hisli N. Emotional state assessment scale that measures the characteristic attitude and depression symptoms. The application takes about 10-15 minutes to complete. It is designed for people aged 13 and over. Scoring and evaluation of scales is easy. The total number of points counted from each four-sentence sentence group is found. For depression scale; 0-9: Normal level, 10-16: Mild depression, 17-29: Moderate depression, 30-63: Indicates severe depression. For anxiety scale; Normal range between 0-7 points, mild anxiety between 8-15 points, middle anxiety between 16-25 points, and severe anxiety between 26-63 points.

ELIGIBILITY:
Inclusion Criteria:

* between 30 and 45 years of age
* who had a tension-type headache diagnosis
* presence of tenderness points on the upper part of the trapezius
* voluntary or written volunteers to participate in the study

Exclusion Criteria:

* cervical area surgery and / or surgery, cervical trauma history
* systemic disease targeting this area
* moderate or excessive nausea and vomiting with headache
* headache due to other causes (e.g., subarachnoid hemorrhage, cerebral hemorrhage, cerebral embolism, cerebral thrombosis, vascular malformation, arthritis, hypertension, or arteriosclerosis)
* have used prophylactic headache medications in the last 3 months
* neurological, mental, hemorrhagic disease, allergy, serious heart, liver, kidney and other organ deficiencies

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Estimated)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-06-10 (Actual); Study Completion 2018-09-25 (Estimated)

PRIMARY OUTCOMES:
Pain thershold | 2 minute
  The algometer is a mechanical pressure device with a minimum diameter of 100 g and a pressure of 10 kg / cm2, with a spring-loaded cylinder with a rubber tip, a circle and a pressure surface of 1 cm2 in diameter, obtained in kg / cm2. Before measuring with the algometer, a pressure of approximately 4 kg was applied to the midpoint of the upper part of the trapezius muscle, which is the control point, with the pulp of the thumb of the hand. Then the force was applied to the same point, causing pain to separate the patient's sense of pressure and pain sensation. This process has been repeated several times. Measurements with an algometer were made at a rate of 1 kg per second. The measurements were interrupted for at least 15-20 seconds. Three measurements were made at these 2 sensitive points and the average of the measurements was recorded.

SECONDARY OUTCOMES:
Pain intensity | 1 minutes
  Visual Analog Scale (VAS) is used to convert some numerical values, such as pain, to numeric values. The two extremes of a 100 mm line are to be assessed on two extremes and the patient is asked to indicate on the line where the severity of the pain is appropriate by drawing a line or placing a point or pointing. The length of the distance from where the pain has never occurred to the point the patient has marked indicates the pain of the patient
Questionnaire | 15 minutes
  Beck Depression Inventory (BDI) and Beck Anxiety Inventory (BAI) developed by Aron T. Beck in 1961, Turkish validity and reliability were done by Hisli N. Emotional state assessment scale that measures the characteristic attitude and depression symptoms. The application takes about 10-15 minutes to complete. It is designed for people aged 13 and over. Scoring and evaluation of scales is easy. The total number of points counted from each four-sentence sentence group is found. For depression scale; 0-9: Normal level, 10-16: Mild depression, 17-29: Moderate depression, 30-63: Indicates severe depression. For anxiety scale; Normal range between 0-7 points, mild anxiety between 8-15 points, middle anxiety between 16-25 points, and severe anxiety between 26-63 points

CONTACTS AND LOCATIONS:
Overall Officials: TOMRIS DUYMAZ, Principal Investigator — Istanbul Bilgi University
Locations (1):
- Tomris Duymaz, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided